CLINICAL TRIAL: NCT04304547
Title: Phase I Clinical Trial to Compare the Pharmacokinetics and Safety of CKD-348 With Co-administration of CKD-828, D097 and D337 in Healthy Adult Volunteers
Brief Title: Clinical Study to Evauate the Pharmacokinetic Profiles and Safety of CKD-348 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A86_04BE1913P
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence A (Active Comparator): CKD-828, D097, D337, CKD-348 T1, CKD-348 T2
  Interventions: Drug: CKD-828, D097, D337, CKD-348 T1, CKD-348 T2
- Sequence B (Active Comparator): CKD-828, D097, D337, CKD-348 T1, CKD-348 T2
  Interventions: Drug: CKD-348 T1, CKD-348 T2, CKD-828, D097, D337,
- Sequence C (Active Comparator): CKD-828, D097, D337, CKD-348 T1, CKD-348 T2
  Interventions: Drug: CKD-348 T2, CKD-348 T1, CKD-828, D097, D337

INTERVENTIONS:
Drug: CKD-828, D097, D337, CKD-348 T1, CKD-348 T2 — Subject of sequence A takes IP in the following order:
  1. Each tablet of CKD-828 and D097 and D337 be taken at once
  2. CKD-348 T1 1 tablet
  3. CKD-348 T2 1 tabet
  Other Names: Sequence A
  Arms: Sequence A
Drug: CKD-348 T1, CKD-348 T2, CKD-828, D097, D337, — Subject of sequence B takes IP in the following order:
  1. CKD-348 T1 1 tablet
  2. CKD-348 T2 1 tablet
  3. Each tablet of CKD-828 and D097 and D337 be taken at once
  Other Names: Sequence B
  Arms: Sequence B
Drug: CKD-348 T2, CKD-348 T1, CKD-828, D097, D337 — Subject of sequence C takes IP in the following order:
  1. CKD-348 T2 1 tablet
  2. Each tablet of CKD-828 and D097 and D337 be taken at once
  3. CKD-348 T1 1 tablet
  Other Names: Sequence C
  Arms: Sequence C

SUMMARY:
Phase I clinical trial to compare the pharmacokinetics and safety of CKD-348 with co-administration of CKD-828, D097 and D337 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. 19 ≤ age ≤ 45
2. Health Volunteers
3. Subject who agreeds to participate in this clinical trial voluntarily

Exclusion Criteria:

1. Subject who cannot participate in a clinical trial based on the PI's judgment

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 hour ~ 144 hr
  Maximum plasma concentration of the drug
AUCt | 0 hour ~ 144 hour
  Area under the concentration time curve from time zero to time

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Chung, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea